CLINICAL TRIAL: NCT01524809
Title: A Single-Centre, Randomised, Double-Blind, 2- Period Crossover Trial Investigating the Steady State Pharmacokinetics of Biphasic Insulin Aspart 30 and Biphasic Insulin Aspart 70 in Subjects With Type 1 Diabetes
Brief Title: Pharmacokinetics of Biphasic Insulin Aspart 30 and 70 in Subjects With Type 1 Diabetes
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: BIASP-1317
Record Dates: First submitted 2012-01-31; First posted 2012-02-02 (Estimated); Last update posted 2017-01-05 (Estimated); Status verified 2017-01

CONDITIONS: Diabetes; Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1 | interventions — insulin aspart, insulin aspart protamine drug combination 30:70

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment period 1 (Experimental)
  Interventions: Drug: biphasic insulin aspart 30; Drug: biphasic insulin aspart 70
- Treatment period 2 (Experimental)
  Interventions: Drug: biphasic insulin aspart 30; Drug: biphasic insulin aspart 70

INTERVENTIONS:
Drug: biphasic insulin aspart 30 — Dose individually adjusted. Administrated subcutaneously (s.c., under the skin) three times a day for 15 days in each treatment period. A wash-out period of 2-8 weeks will take place between treatment periods.
Drug: biphasic insulin aspart 70 — Dose individually adjusted. Administrated subcutaneously (s.c., under the skin) three times a day for 15 days in each treatment period. A wash-out period of 2-8 weeks will take place between treatment periods.

SUMMARY:
This trial is conducted in Europe. The aim of this trial is to investigate steady state pharmacokinetics of biphasic insulin aspart 30 and biphasic insulin aspart 70 in subjects with type 1 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetes for at least 12 months
* Currently on a multiple dose insulin regimen
* HbA1c maximum 12.0%
* BMI (body mass index) below 35 kg/m^2
* Able and willing to perform self-blood glucose monitoring (SBGM)

Exclusion Criteria:

* Treatment with insulin aspart within the last 14 days prior to this trial
* The receipt of any investigational drug within the last 30 days prior to this trial
* Total daily insulin dose at least 1.8 U/kg
* A history of drug abuse or alcohol dependence within the last 5 years
* Impaired hepatic function
* Impaired renal function
* Blood donation within the last nine weeks or haemoglobin below the lower reference limit according to the local laboratory
* Cardiac disease
* Severe, uncontrolled hypertension

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2001-01; Primary Completion 2001-06 (Actual); Study Completion 2001-06 (Actual)

PRIMARY OUTCOMES:
Area under the serum insulin curve 6-14 hours after dinner at day 15

SECONDARY OUTCOMES:
Area under the serum insulin curve 6-14 hours after dinner at day 1
Area under the serum insulin curve 0-6 hours after dinner
Area under the curve 0-24 hours
Serum insulin
Apparent t½ (apparent elimination half life)
Cmax, maximum concentration
tmax, time to reach Cmax
Adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR,1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Århus C, Denmark

REFERENCES:
- [Result] Chen JW, Lauritzen T, Christiansen JJ, Jensen LH, Clausen WH, Christiansen JS. Pharmacokinetic profiles of biphasic insulin aspart 30/70 and 70/30 in patients with Type 1 diabetes: a randomized double-blinded crossover study. Diabet Med. 2005 Mar;22(3):273-7. doi: 10.1111/j.1464-5491.2004.01404.x. PMID 15717874
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com